CLINICAL TRIAL: NCT07096635
Title: Effect of Preoperative Oral Melatonin With Intra Articular Analgesia on Post-Operative Pain Relief After Arthroscopic Anterior Cruciate Ligament Reconstruction Under Spinal Anesthesia. A Randomized Comparative Controlled Clinical Trial
Brief Title: Oral Melatonin With Intra Articular Analgesia on Pain After Arthroscopic Anterior Cruciate Ligament Reconstruction
Acronym: ACLR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seham Mohamed Moeen Ibrahim, Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SM72025
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Pain Relief After Arthroscopic Anterior Cruciate Ligament Reconstruction
MeSH Terms: interventions — Melatonin; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M (Active Comparator): Patients will receive oral melatonin 10 mg (two 5 mg tablets) one hour before the operation plus intra-articular analgesia at the end of surgery.
  Interventions: Drug: Melatonin
- Group C (Placebo Comparator): Patients will receive two oral inert starch tablets of the same shape and color one hour before the operation plus intra-articular analgesia at the end of surgery.
  Interventions: Other: Starch tablets

INTERVENTIONS:
Drug: Melatonin — Patients will receive oral melatonin 10 mg (two 5 mg tablets) one hour before the operation plus intra-articular analgesia at the end of surgery.
  Arms: Group M
Other: Starch tablets — Patients will receive two oral inert starch tablets of the same shape and color one hour before the operation plus intra-articular analgesia at the end of surgery.
  Arms: Group C

SUMMARY:
Anterior Cruciate Ligament Reconstruction (ACLR) is a common orthopedic procedure that is accompanied by moderate to severe postoperative pain and is primarily performed on an outpatient basis.

DETAILED DESCRIPTION:
Many different pain control treatments are used in the management of patients after ACLR, including various permutations of nerve blocks, nerve block adjuncts (NBAs), intra-articular injections, intravenous (IV), oral medications, and cryotherapy, as well as compression stockings. Despite this, no gold-standard postoperative analgesia guideline has emerged.

Melatonin (N-acetyl-5-methoxytryptamine) is a naturally-occurring hormone in the human body and offers antiemetic, analgesic, and anxiolytic effects

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective unilateral arthroscopic reconstruction of the anterior cruciate ligament (ACL) under spinal anesthesia, aged from 18 to 65 years old, and who are American Society of Anesthesiologists (ASA) physical status I or II of either sex

Exclusion Criteria:

* Contraindications to neuraxial anesthesia (e.g. allergy to local anesthetics, coagulopathies, infection in the area)
* History of cardiovascular, cerebrovascular, respiratory, or psychological disorders
* Chronic pain syndrome and/ or opioid use
* Regular consumption of analgesics, corticosteroids or anticonvulsants
* A known allergy to melatonin
* Patients with diabetes mellitus, sever hypertension, liver or renal dysfunction
* Cognitive disorders (dementia, major depression)
* Circadian rhythm disorders (such as chronic fatigue syndrome and drowsiness)
* Pregnancy/ lactating
* Body mass index 35 kg/m2 or more,
* Patient refusal.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Time to first analgesic requirement | 24 hours after surgery
  Assessed in minutes

SECONDARY OUTCOMES:
Postoperative pain intensity | 24 hours after surgery
  Assessed by the visual analogue scale, an 11-point scale graded from 0 to 10 (0 = no pain, 10 = the worst imaginable pain)

CONTACTS AND LOCATIONS:
Overall Officials: Seham M Moeen, M.D., Principal Investigator — Assiut University